CLINICAL TRIAL: NCT03435549
Title: Automated Hovering for Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 828882
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Joint Disease
MeSH Terms: conditions — Joint Diseases | interventions — Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Control Arm (Usual care) (No Intervention): If Patient is randomized to Arm 1, no contact will occur, patient will receive standard and routine clinical care
- Arm 2a: Remote monitoring (Experimental): If Patient is randomized to Arm 2a they will remote monitoring for 6 weeks post-surgery
  Interventions: Behavioral: Remote monitoring
- Arm 2b: Remote monitoring plus goal setting and social support (Experimental): If Patient is randomized to Arm 2b, they will receive a remote monitoring plus social support and nudge messaging for 6 weeks post-surgery
  Interventions: Behavioral: Remote monitoring plus goal setting and social support

INTERVENTIONS:
Behavioral: Remote monitoring — Patients given an activity tracker to wear for 6 weeks after LEJR replacement surgery. For 2 weeks after surgery, they will also receive a daily text messages asking what their pain is on a scale of 0 to 10. They will be asked to reply to the text with their pain score. They will also be sent occasional messaging about their recovery, tips of what to do, and feedback on their progress. They will also also be sent a text message if they stop using their activity tracker for 3 days.
  Arms: Arm 2a: Remote monitoring
Behavioral: Remote monitoring plus goal setting and social support — Patients given activity tracker to wear for 6 weeks after LEJR surgery. For 2 weeks after surgery, they will receive a daily text messages asking what their pain is on a scale of 0 to 10 and asked to reply by text. They will be sent occasional messaging about their recovery, tips of what to do, and feedback on their progress. They will also also be sent a text message if they stop using their activity tracker for 3 days. Patients will be asked to identify a a friend or family member to act as support partner. The study will share progress updates with support partner and contact this individual if patient stops wearing the activity tracker for over 3 days. This partner will also be able to provide supportive messages to help encourage them to reach their activity goals.
  Arms: Arm 2b: Remote monitoring plus goal setting and social support

SUMMARY:
This will evaluate the effectiveness of automated hovering to encourage patients to be discharged to home after hip or knee replacement surgery. Automated hovering includes monitoring of physical activity with an activity monitor, tracking of pain scores, daily feedback and motivational messages, social influence, and connection to clinicians as needed.

DETAILED DESCRIPTION:
The goal of this study is to test the approach of automated hovering to encourage patients to be discharged to home safely after lower extremity joint replacement surgery (LEJR). The investigators will target those patients undergoing hip or knee replacement surgery at a large urban hospital system at two different sites. The investigators aim is to increase the number of patients that are discharged to home, by providing patients with a physical activity pedometer, daily pain score tracking through bi-directional text messaging, milestone and nudge messaging for recovery, social influence, and connection to clinicians as needed for 6 weeks after surgery. Eligible participants are age 18-85, with a Risk Assessment and Prediction Tool (RAPT) score of 6-8 and are scheduled to undergo lower-extremity joint replacement surgery. Participants will be randomized 1:1 to usual care (Arm 1) and intervention (Arms 2a and 2b). After enrollment with the monitoring device, participants in the intervention group will be randomized 1:1 to Arm 2a (remote monitoring) or Arm 2b (remote monitoring + goal-setting and social support). Both intervention arms will receive the intervention for 6 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria: University of Pennsylvania Health System (UPHS) patients between the ages of 18-85 with a Risk Assessment and Prediction Tool (RAPT) of 6-8 and scheduled to undergo primary lower-extremity joint replacement surgery.

Exclusion Criteria:

* Patients will be excluded if they do not meet all of the inclusion criteria, or if they have bilateral or revision surgery, dementia, end stage renal disease, cirrhosis, metastatic cancer, non- English speaker, or other physical impairment (ex. amputation)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Discharged to home | Day of discharge through study completion at 6 weeks
  % of patients discharged to home
Step increase | 6 weeks post discharge
  % of step increase as measured by activity tracker

SECONDARY OUTCOMES:
Days spent at home | 6 weeks post discharge
  Number of days spent at home after discharge
Timed Up and Go (TUG) score | 6 weeks post discharge
  % change in TUG score

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Hume E, Troxel AB, Reitz C, Norton L, Lacko H, McDonald C, Freeman J, Marcus N, Volpp KG, Asch DA. Effect of Remote Monitoring on Discharge to Home, Return to Activity, and Rehospitalization After Hip and Knee Arthroplasty: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2028328. doi: 10.1001/jamanetworkopen.2020.28328. PMID 33346847